CLINICAL TRIAL: NCT03927872
Title: Cardio-embolic Stroke and Blood Bio-markers:Diagnosis and Predictors of Short Term Outcome.
Brief Title: Cardio-embolic Stroke and Blood Bio-markers
Status: Completed | Type: Observational
Sponsor: Wafaa Samir (Other Government)
Responsible Party: Sponsor-Investigator, Wafaa Samir, Assistant professor of neurology, Zagazig University
Organization: Zagazig University (Other Government)
Other Study IDs: ZU-IRB# :2325/7-9-2015).
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cardioembolic stroke
  Interventions: Other: blood biomarkers
- non cardioembolic stroke
  Interventions: Other: blood biomarkers

INTERVENTIONS:
Other: blood biomarkers — assessment of serum BNP, D-Dimer and CK-MB and CRP and globulin /albumin ratio stroke outcome

SUMMARY:
Brain is a productive source of variety of enzymes and any brain injury like stroke to brain tissue could similarly result in an increase in these enzymes in cerebrospinal fluid and serum. Evaluation of these enzymes represent a simple method for the ischemic stroke subtype diagnosis and prognosis .Objective: The aim of this study was to determine the role Brain natriuretic peptide (BNP) , D-Dimer , creatine kinase- MB(CK-MB) , C reactive protein (CRP) serum levels and G/A ratio in diagnosis of CES stroke and its ability to predict short term outcome. Methods: This study was conducted on 96 patients with acute ischemic stroke, subdivided into two groups, group Ι was 48 patients with cardio-embolic stroke and group ΙΙ was 48 patients with non- cardio-embolic. all patients were subjected to assessment of serum BNP, D-Dimer and CK-MB and CRP and globulin /albumin ratio within the first 24 h of stroke .At third week ,they were assessed by mRS.

DETAILED DESCRIPTION:
participants and methods : 96 acute ischemic stroke patients divided to two groups ; group Ι : 48 patients with cardio-embolic stroke (CES) and group ΙΙ: 48 patients with cerebrovascular stroke other than cardio-embolic stroke (non CES), with first-ever acute ischemic stroke within 24 h of onset of symptoms admitted to Intensive Care and Stroke Unit .

All patients were subjected to full detailed neurological history with stressing on the vascular and cardiac risk factors , and general and neurological examination. Stroke severity was assessed using Glasgow Coma Scale (GCS) and the National Institutes of Health Stroke Scale (NIHSS)

Laboratory investigations:15 ml venous blood were obtained from the patients within the first 24 hours of stroke. All routine and special laboratory investigations were done at Clinical pathology department, Zagazig university hospitals including CBC, liver function, kidney function, ESR and lipid profile.

Brain natriuretic peptide : 4 ml blood was placed in a polypro pane tube containing a mixture of sodium salt of ethylene diamine tetra acetic acid (EDTA) at a concentration of 1mg /ml of blood and aprotinin at a concentration of 500 kallikerin inhibitory unit (kiu) /ml of blood serving as a natural proteinase inhibitor which act as a preservative for natriuretic peptides , then mixing of the blood was done . then the tube was centrifuged at 5000 rpm for 15 minutes in the cool centrifuge , the separated serum was stored at -70 degree c until analysis.

Later on the assay was done using human BNP Elisa kits (Spain react kits sr 19369u) which are immune-sorbent assay for quantitative measurement , the least sensitivity is 14 pg/ml and ranges 14 -1000pg/ml .

D-Dimer: 3ml blood was collected within a vacuum tubes containing 0.5 ml buffered sodium citrate before the initiation of any oral, enteral or parenteral feeding or medications. Blood samples were mixed well with avoiding of foam formation then immediately centrifuged at 3000 rpm for 15 min at ambient room temperature and plasma is separated. D-Dimer was measured turbidmetry (SAT Liatest D-Di; Diagnostica STAGO) on the STAgo compact analyzer, Normal value is less than 500 ng / ml (15).

Creatine Kinase MB : 4 ml blood were derived within a plastic tube centrifuged at 4000rpm for 3minutes , the separated serum was assayed for CK MB using Spain react kits with normal value up to 2.8ng /L C reactive protein : 4ml were withdrawn in a plastic tube centrifuged at 4000rpm for 3minutes , the separated serum used for analysis of CRP measured using Olympus 640 analyzer with normal value up to 5 mg / L Globulin/Albumin ratio( G/A) was calculated with normal ratio 0.6-0.7 . All patients were evaluated by Brain CT or MRI for diagnosis of ischemic stroke .

Each patient underwent to Electrocardiogram, Echocardiography and Carotid Doppler ultrasonography to define etiological stoke subtype.

ELIGIBILITY:
Inclusion criteria:

* CES and non- CES diagnosis was according to Trial of Org 10172 in Acute Stroke Treatment ﴾TOAST﴿ classification criteria.
* non -CES were selected to match patients with CES regarding age and vascular risk factors as a control group.
* Patients with National Institutes of Health Stroke Scale ﴾NIHSS ﴿ score more than 5.
* Adult patients with their ages more than 18 year.

Exclusion criteria:

* Lacunar stroke and transient ischemic attacks (TIAs)
* Haemorrhagic stroke.
* Neurological causes of acute focal cerebral dysfunction such as cerebral venous sinus thrombosis , head trauma, infection, and auto immune disorders
* Heart failure
* Liver failure
* Chronic renal disease.

Ages: 32 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 96 AIS patients divided to two groups ; group Ι : 48 patients with cardio-embolic stroke (CES) and group ΙΙ: 48 patients with cerebrovascular stroke other than cardio-embolic stroke (non CES), with first-ever acute ischemic stroke within 24 h of onset of symptoms admitted to Intensive Care and Stroke Unit
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
modified rankin scale | at the third week of stroke onset
  ranging from zero(no symptoms at all) to 6 (dead).outcome was defined as good if mRS=0-2,bad (poor) if mRS=3-5 and death if mRS=6

IPD SHARING:
Plan to Share IPD: No